CLINICAL TRIAL: NCT05853432
Title: A Descriptive Study of Baseline Characteristics, Clinical Outcomes, and Treatment Patterns of HR+/HER2- Advanced or Metastatic Breast Cancer Patients Treated With Alpelisib Plus Fulvestrant Who Have Received Fulvestrant in Any Prior Line of Therapy
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBYL719C2009
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: HR+/HER2- Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This was a non-interventional, retrospective cohort study of patients with HR+/HER2- aBC treated with alpelisib (ALP) plus fulvestrant (FUL) who have received fulvestrant in any prior line of therapy (LoT). This study utilized de-identified individual patient data from the United States (US) ConcertAI Patient360 Breast Cancer database, sourced from electronic health records (EHR) (i.e., secondary use of data). Patients were indexed at their start date of the earliest alpelisib plus fulvestrant regimen and followed until their death date or last confirmed activity date in the absence of an observed death.

ELIGIBILITY:
Inclusion Criteria:

* Had a curated record for advanced or metastatic breast cancer diagnosis.
* Note: Diagnosis of a/mBC is based on a curated record of M stage=M1, Stage 4/4a/4b, presence of metastatic tumor, Stage 3b/3c or presence of secondary neoplasm.
* Had patient activity documented in ConcertAI Patient 360 Breast Cancer database (defined as a record of a clinic visit, medication administration, vital test, or lab test) or death within 90 days after the advanced or metastatic breast cancer diagnosis date.
* Had documented receipt of treatment with alpelisib plus fulvestrant on or after the advanced or metastatic diagnosis date.
* Had documented receipt of treatment with fulvestrant before the index date (start date of the earliest alpelisib plus fulvestrant regimen). This included (neo) adjuvant therapies.
* Age ≥18 years on the index date.

Exclusion Criteria:

* Had documented hormone receptor-negative (defined as both estrogen receptor-negative and progesterone receptor-negative) or HER2-positive status any time prior to index date (but prioritizing results closest to index date, if there were conflicting results).
* Patient had a clinical trial registration date (i.e., participated in a clinical trial) on or before the index date.
* Patients with "negative" PIK3CA test before index date (in case of multiple tests, the one closer to the index date was used).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to approximately 21 months
  OS was defined as the length of time from the start date of the earliest alpelisib plus fulvestrant regimen to the date of death, or last confirmed activity date in the absence of an observed death event.
Real-world progression-free survival (rwPFS) | Up to approximately 21 months
  rwPFS was defined as the length of time from the start date of the earliest alpelisib plus fulvestrant regimen to the first documented progression or death date occurring at least 14 days after the index date, or last adequate tumor assessment date in the absence of an observed progression or death event.
Line of treatment of ALP+FUL received | Baseline
Line of treatment number of index regimens stratified by index year | Baseline
Starting dose of alpelisib | Baseline
Number of prior regimens | Baseline
Prior fulvestrant treatment category | Baseline
Prior regimens of patients who received alpelisib plus fulvestrant as first-line treatment | Baseline
Number of prior fulvestrant regimens prior to alpelisib plus fulvestrant | Baseline
Percentage of patients with prior exposure to CDK4/6i in the adjuvant setting | Baseline
Percentage of patients with prior exposure to chemotherapy in the metastatic setting | Baseline
Time to treatment discontinuation | Up to approximately 21 months
First antineoplastic regimen received after discontinuation of the alpelisib plus fulvestrant regimen | Up to approximately 21 months

SECONDARY OUTCOMES:
Overall survival (OS) in subgroups of patients according to the prior lines of treatment | Up to approximately 21 months
  OS was defined as the length of time from the start date of the earliest alpelisib plus fulvestrant regimen to the date of death, or last confirmed activity date in the absence of an observed death event.
Real-world progression-free survival (rwPFS) in subgroups of patients according to the prior lines of treatment | Up to approximately 21 months
  rwPFS was defined as the length of time from the start date of the earliest alpelisib plus fulvestrant regimen to the first documented progression or death date occurring at least 14 days after the index date, or last adequate tumor assessment date in the absence of an observed progression or death event.
Line of treatment of ALP+FUL received in subgroups of patients according to the prior lines of treatment | Baseline
Line of treatment number of index regimens stratified by index year in subgroups of patients according to the prior lines of treatment | Baseline
Starting dose of alpelisib in subgroups of patients according to the prior lines of treatment | Baseline
Number of prior regimens in subgroups of patients according to the prior lines of treatment | Baseline
Prior fulvestrant treatment category in subgroups of patients according to the prior lines of treatment | Baseline
Prior regimens of patients who received alpelisib plus fulvestrant as first-line treatment in subgroups of patients according to the prior lines of treatment | Baseline
Number of prior fulvestrant regimens prior to alpelisib plus fulvestrant in subgroups of patients according to the prior lines of treatment | Baseline
Percentage of patients with prior exposure to CDK4/6i in the adjuvant setting in subgroups of patients according to the prior lines of treatment | Baseline
Percentage of patients with prior exposure to chemotherapy in the metastatic setting in subgroups of patients according to the prior lines of treatment | Baseline
Time to treatment discontinuation in subgroups of patients according to the prior lines of treatment | Up to approximately 21 months
First antineoplastic regimen received after discontinuation of the alpelisib plus fulvestrant regimen in subgroups of patients according to the prior lines of treatment | Up to approximately 21 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Dublin, Ireland